CLINICAL TRIAL: NCT00010985
Title: Usual Care Vs Choice of Alternative Rx: Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01 AT000144-01M; R01AT000144-01 (NIH); NCT00008918 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Acute Low Back Pain
Keywords: Backpain; Pain; Alternative Medicine; Acupuncture; Chiropractic; Massage Therapy
MeSH Terms: conditions — Back Pain; Pain | interventions — Acupuncture Therapy; Manipulation, Chiropractic; Massage

INTERVENTIONS:
Procedure: Acupuncture
Procedure: Chiropractic
Procedure: massage

SUMMARY:
This study compares two approaches to the management of acute low back pain: usual care (standard benefit) vs. the choice of: usual care, chiropractic, acupuncture or massage therapy (expanded benefit). 480 subjects with uncomplicated, acute low back pain will be recruited from a health maintenance organization, and randomized to either usual care (n=160) or choice of expanded benefits (n=320). Patients' preferences for individual therapies and expectations of improvement will be measured at baseline and throughout the study. Subjects randomized to the expanded benefits arm who choose chiropractic, acupuncture or massage will receive up to 10 treatments over a five-week period. Additional treatments will be available after the fifth week but will require a copayment. Treatments will be provided by licensed providers who have met strict credentialing criteria. Chiropractic, acupuncture or massage treatments will begin within 48 hours. Chiropractic, acupuncture and massage therapy scope of practice guidelines for the treatment of acute low back pain have been developed as have detailed data tracking procedures to be used at each patient visit. Symptom relief, functional status, restricted activity days, use of health care, and patient and provider satisfaction will be assessed at 2, 5,12, 26 and 52 weeks after initiation of treatment. Primary outcomes will include: 1) change in symptoms; 2) change in functional status; 3) patient satisfaction; and 4) total utilization of services associated with care for low back pain. Medical records and the HMO's cost management information system will identify use of services. It is hypothesized that patients offered their choice of expanded benefits will experience a more rapid improvement in symptoms, a faster return to baseline functional status, a decrease in utilization of conventional medical services, and will be more satisfied with their care. The study is a direct examination of the effectiveness of an insurance eligibility intervention, not a test of the efficacy of specific, non-allopathic treatment regimens. The results of this study will provide valuable information to clinicians, patients and third party payers on the relative benefits and costs of an "expanded benefits" treatment option which incorporates chiropractic, acupuncture and massage services for low back pain.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* Backpain for less than 21 days
* Backpain within the last 24 hours
* No prior treatment or evaluation for this episode of backpain
* Ability to read and speak English

Exclusion Criteria:

* Not low backpain
* Backpain for >21 days
* Already evaluated for this episode of backpain
* Already treated with acupuncture, chiropractic, massage therapy, or physical therapy for this episode of backpain
* Osteoporosis
* Taking systemic corticosteroids
* Pregnancy
* History of cancer (other than non-melanoma skin cancer)
* Clotting disorders or currently taking anti-coagulant medication
* Severe or disabling co-exiting problem (e.g. fibromyalgia, substance abuse, rheumatoid arthritis, etc.)
* Unable to read or speak English
* History of back or neck surgery within the last 5 years
* History of vertebral fracture or dislocation
* Neurological symptoms suggestive of Cauda Equina Syndrome
* Requires immediate referral to specialist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: David Eisenberg, MD, Principal Investigator — Harvard Medical School Osher Institute
Locations (1):
- Harvard Medical School Osher Institute, Boston, Massachusetts, United States